CLINICAL TRIAL: NCT04055506
Title: An Open-label, Single-sequence Study to Investigate the Effects of Cytochrome P450 1A2 Induction by Ritonavir on the Pharmacokinetics of BMS-986165 in Healthy Participants
Brief Title: A Study to Investigate the Effects of Cytochrome P450 1A2 Induction by Ritonavir on BMS-986165 Drug Levels and Effects in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IM011-087
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — deucravacitinib; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental)
  Interventions: Drug: BMS-986165; Drug: Ritonavir

INTERVENTIONS:
Drug: BMS-986165 — Dose 1
Drug: Ritonavir — 100 mg

SUMMARY:
The Study of Cytochrome P450 1A2 Induction by Ritonavir on the drug effects of BMS-986165 in Healthy Participants

ELIGIBILITY:
Inclusion Criteria:

* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) > 80 mL/min/1.732 m2 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic onadotropin) within 24 hours prior to the start of study treatment.
* Body mass index of 18.0 kg/m2 to 32.0 kg/m2, inclusive, and body weight ≥ 50 kg, at screening.

Exclusion Criteria:

* Participants who currently smoke, as well as those who have stopped smoking less than 6 months prior to dosing on Day 1.
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population.
* Prisoners or participants who are involuntarily incarcerated
* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986165 | Day 1
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration of BMS-986165 | Day 1
Area under the plasma concentration-time curve from time zero extrapolated to infinite time in BMS-986165 | Day 1
Maximum observed plasma concentration of BMS-986165 in combination with steady-state ritonavir | Day 15
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration of BMS-986165 in combination with steady-state ritonavir | Day 15
Area under the plasma concentration-time curve from time zero extrapolated to infinite time in BMS-986165 in combination with steady-state ritonavir | Day 15

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | initial dose up to day 29
vital signs of blood pressure | initial dose up to day 29
Vital signs of body temperature | initial dose up to day 29
Vital signs of respiratory rate | initial dose up to day 29
Number of Clinically significant changes in lab assessment of blood serum | initial dose up to day 29
Number of Clinically significant changes in the lab assessment of blood | initial dose up to day 29
Number of Clinically significant changes in the lab assessment of urine | initial dose up to day 29

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm